CLINICAL TRIAL: NCT07119333
Title: Classroom Air Purifiers for Reducing School Absence: Protocol for a Cluster-randomized, Parallel, Two-arm, Group Sequential Superiority Trial
Brief Title: Classroom Air Purifiers for Reducing School Absence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 737650
Record Dates: First submitted 2025-08-11; First posted 2025-08-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Asenteeism
Keywords: Randomized trial; Air purifiers; Student absenteeism; respiratory infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Air Filters

STUDY DESIGN:
Intervention Model Description: The intervention is the installation and operation of two portable air purifiers with HEPA filters per intervention school classroom. Each air purifier will operate at a level corresponding to 3.0 air changes per hour, providing a combined capacity corresponding to a Clean Air Delivery Rate (CADR) of at least 486 m3/hour.
  The control is the installation and operation of two sham air purifiers per control classroom. These will be identical in appearance and placement to the intervention units and will also include a HEPA filter, but they will be modified by the manufacturer to operate at the lowest fan setting permitted by the motor. This setting results in minimal airflow and negligible air-cleaning capacity but may also produce less sound than the intervention units. The sham air purifiers will operate at a performance equivalent to 0.3 air changes per hour, providing a combined CARD of at least 48 m3/hour
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: School staff, participating teachers, and students will be blinded to treatment allocation via the use of sham air purifiers in the control group. The researchers responsible for installing the air purifiers will also be blinded. To ensure this, all air purifier units will be configured and labeled with serial numbers indicating whether they are sham or functional devices, with one identifier placed in a clearly visible location and another in an inaccessible location. Prior to installing, the visible identifier will be replaced with a label displaying the school and classroom names according to an allocation key, which will be securely stored and accessible only to a single designated researcher (SH). This researcher will configure the air purifiers assigned to the control and intervention arms and will be the sole individual with knowledge of treatment allocation until the point of unblinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is the installation and operation of two portable air purifiers with HEPA filters per intervention school classroom. Each air purifier will operate at a level corresponding to 3.0 air changes per hour, providing a combined capacity corresponding to a Clean Air Delivery Rate (CADR) of at least 486 m3/hour.
  Interventions: Device: Air purifiers
- Control (Sham Comparator): The control is the installation and operation of two sham air purifiers per control classroom. These will be identical in appearance and placement to the intervention units and will also include a HEPA filter, but they will be modified by the manufacturer to operate at the lowest fan setting permitted by the motor. This setting results in minimal airflow and negligible air-cleaning capacity but may also produce less sound than the intervention units. The sham air purifiers will operate at a performance equivalent to 0.3 air changes per hour, providing a combined CARD of at least 48 m3/hour.
  Interventions: Device: Sham air purifiers

INTERVENTIONS:
Device: Air purifiers — Air purifiers
  Arms: Intervention
Device: Sham air purifiers — Sham air purifiers
  Arms: Control

SUMMARY:
Background

Respiratory infections like influenza and SARS-CoV-2 pose significant global health risks due to their high transmissibility and severity. SARS-CoV-2 has caused over 7 million deaths worldwide, and the Lancet Commission estimates a >20% chance of a similar respiratory virus pandemic within a decade. Schools, often poorly ventilated, are high-risk settings for transmission. While COVID-19 school closures may have reduced transmission, they likely caused learning loss, mental health issues, and increased burdens on parents and caregivers. Air purifiers with HEPA filters may offer a non-disruptive mitigation strategy, but the evidence to support their effectiveness in reducing viral transmission is weak. This protocol describes a cluster-randomised, parallel, two-arm, group sequential superiority trial with an interim analysis-to allow early stopping for efficacy or futility-to estimate the effect of portable air purifiers with HEPA filters in primary school classrooms on student absenteeism.

Research Questions

The primary question is whether installing and operating air purifiers with HEPA-filters (intervention) reduce student absenteeism (primary outcome) compared to sham air purifiers (control). Secondary questions examine whether the intervention reduces teacher absenteeism due to respiratory infections, rate and 12-week risk of self-reported respiratory infections among teachers, and teachers' perceived air quality compared to sham air purifiers. If the trial estimates a statistically significant effect for the primary outcome, a cost-consequence analysis will evaluate the direct and indirect costs associating with operating air purifiers against the potential benefits of reduced student and teacher absenteeism. A process evaluation will explore mechanisms of effect.

Methods and Analysis

This group sequential trial will randomize schools (clusters) 1:1 to intervention or control arms in two stages: winter 2025/2026 (N = 32 schools; ~736 students) and winter 2026/2027 (N = 30 schools; ~690 students). Eligible schools must have classrooms suitable for portable air purifiers, >10 students in grades 5-7 (typically aged 10-13 years), and principal consent. Intervention and control classrooms will each receive two portable air purifiers with HEPA-filters operating at a performance equivalent to 3.0 and 0.3 air changes per hour, respectively, with control purifiers acting as shams.

Outcomes will be measured during and at the end of a 12-week period. The primary outcome is student absenteeism, measured as full child-days of absence aggregated at the class level. An interim analysis is planned at the end of the first stage, with error-spending O'Brien-Fleming stopping boundaries that are binding for efficacy and nonbinding for futility.

The primary estimand is the marginal incidence rate ratio of student absences, estimated using generalized estimating equations with a negative binomial model to account for overdispersion. Prespecified stopping boundaries will determine stopping, with efficacy boundaries being binding. Treatment effects will be estimated using cluster-bootstrapped confidence intervals adjusted to provide strong control on overall type I and II error probabilities, and a bias correction will be applied if the trial is stopped early for efficacy. All analyses will follow the intention-to-treat principle.

Ethics and Dissemination

The trial has been approved by the Regional Committees for Medical and Health Research Ethics and the National Research Ethics Committee. Results will be disseminated to stakeholders, participants and the public through peer-reviewed journals, scientific meetings and social media.

ELIGIBILITY:
There are two general trial populations. The first population is primary school children in Norway. Primary school children in primary schools meeting the following criteria will be eligible:

1. Schools with more than 10 students in either 5th, 6th, or 7th grade (typically aged 10-13 years).
2. Schools with at least one classroom of sufficient dimensions to accommodate the installation of two portable air purifiers.
3. The school principal accepts the installation of air purifiers in at least one classroom in the 5th, 6th, or 7th grade that meets the first two inclusion criteria.

For logistical and administrative reasons, the investigators will try to limit the sampling frame to schools in municipalities located close our offices in Oslo. These municipalities include several large towns with populations of around 30 000 to 100 000 people, as well as sparsely populated rural areas, and are therefore reasonably representative of Norway and many other countries. The investigators will enlarge the sampling frame as necessary.

The second population is teachers at primary schools in Norway. Teachers meeting the following criteria will be eligible.

1. Be the main class teacher of one or more of the classrooms included in the trial.
2. Provide informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Student absenteeism | From enrollment to the end of intervention at 12 weeks
  The primary outcome is the number of student-days of absence per classroom, measured each week. The investigators will define a student day of absence as a day for which a student is absent for the entire day. The investigators will not distinguish between the specific students who are absent (i.e., two days of absence will be counted for one student who is absent on two days, and for two students absent for one day each).

SECONDARY OUTCOMES:
Self-reported absence due to respiratory infections among teachers | From enrollment to the end of intervention at 12 weeks
  The investigators will measure the number of teacher-days of work absence (sick leave) due to self-reported respiratory infection each week. The investigators will ask teachers "Did you experience symptoms of a cold, COVID-19 or the flu last week?". Teachers who answer "Yes" to this question, will be asked to specify the symptoms they experienced (sneezing, nasal obstruction, nasal discharge, sore throath, cough, headache, fever or general discomfort) and rate each symptom from 0 to 3, where 0 = absent, 1 = mild, 2 = moderate, 3 = severe, in accordance with the Jackson index. They will then report the number of days they experienced these symptoms (ranging from 1 to 7 days), before answering "How many days were you absent from work last week due to respiratory infection?"; their response to this question will be used to measure number of days of absence. A count of zero days will be assigned to teachers answering "No" to the first question.
Incidence of self-reported respiratory symptoms consistent with respiratory infections among teachers | From enrollment to the end of the intervention at 12 weeks
  The investigators will assess incidents of respiratory symptoms consistent with respiratory infections among teachers using self-reported data collected weekly. The investigators define an incident as a period during which a teacher reports symptoms for at least two consecutive calendar days, preceded and followed by at least 7 symptom-free calendar days. The investigators define symptoms of respiratory infection as meeting all four of the following criteria:
  1. Answering "yes" to the question "Did you experience symptoms of a cold, COVID-19 or the flu last week?".
  2. Reporting at least one of the following symptoms: nasal obstruction (plugged or congested), nasal discharge (runny nose), sneezing or sore throat, in the last week;
  3. Scoring at least four points on the Jackson scale (as assessed for the preceding week);
  4. Reporting that they have experienced at least one of the reported symptoms for at least two consecutive days in the last week.
Teachers reporting respiratory infections | From enrollment to the end of the intervention at 12 weeks
  The investigators will assess respiratory infection as a dichotomous outcome for each teacher, based on whether they meet the case definition at any point during the 12-week follow-up.
Teacher perceptions of air quality in classrooms | From enrollment to the end of the intervention at 12 weeks
  The investigators will assess teachers' perceptions of classroom air quality at the end of follow-up using the MM040 questionnaire: teachers will report whether they have experienced drafts, high room temperature, low room temperature, fluctuating room temperature, stuffy or "bad" air, dry air, unpleasant odours, noise, or dust in the air during follow-up. The response options will be: "Yes, often (every week)," "Yes, occasionally," or "No, never".
Adverse events | From enrollment to the end of the intervention at 12 weeks
  The investigators define an adverse event as any significant disruption to lessons, or any accident or injury, that is attributable to the intervention or control. The investigators will instruct school principals and teachers to report such events.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Institute of Public Health, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes
The final anonymised dataset and statistical code will be archived and made freely available to the public on GitHub and will be assigned a digital object identifier in the main article.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Solberg RB, Holos SB, Elgersma IH, Elstrom P, Rose CJ, Helleve A, Gopinathan U, Fretheim A. Classroom air purifiers for reducing school absence: study protocol for a pragmatic, cluster-randomised, parallel, two-arm, group sequential superiority trial. BMJ Open. 2025 Dec 24;15(12):e109659. doi: 10.1136/bmjopen-2025-109659. PMID 41448709